CLINICAL TRIAL: NCT02806544
Title: Neoadjuvant Endocrine Therapy in Locally Advanced Hormone Receptor Positive Breast Cancer in a Low-Resource, Middle-Income Setting (Guatemala)
Brief Title: Neoadjuvant Tamoxifen in Locally Advanced Breast Cancer in a Low/Middle Income Country
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Washington University School of Medicine (Other); Instituto National de Cancerologia, Guatemala (Unknown)
Responsible Party: Principal Investigator, Laila Saied, Clinical Fellow, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150045
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Results first posted 2016-11-17 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: Breast neoplasms; Breast cancer; Locally advanced breast cancer; Neoadjuvant endocrine therapy; Tamoxifen; Low and middle income country
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tamoxifen (Experimental): Tamoxifen 20mg by mouth daily
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — Tamoxifen 20mg by mouth daily

SUMMARY:
This study evaluates the feasibility and efficacy of neoadjuvant tamoxifen for patients with locally advanced hormone receptor positive breast cancer in a low/middle income country.

DETAILED DESCRIPTION:
This is a single arm feasibility study of neoadjuvant tamoxifen for locally advanced hormone receptor positive breast cancer in a low-resource setting in a middle-income country (Guatemala). Patients will be treated with tamoxifen for four to six weeks, then have an on-treatment biopsy to assess Ki-67. If Ki-67 is less than or equal to 10%, the patient will continue on tamoxifen for a total of 4 months; if Ki-67 is greater than 10% or there is clinical progression, patients will be taken off study. The study will evaluate the proportion of patients treated with four months of tamoxifen who undergo definitive surgery and the clinical and pathologic response rates.

ELIGIBILITY:
Inclusion Criteria:

* Patient evaluated and treated at INCAN
* Patients must provide informed consent
* Patient must be ≥ 18 years of age.
* Life expectancy ≥ 6 months
* Clinical locally advance breast cancer (Stage IIB or III)
* Pathologically confirmed diagnosis of estrogen receptor (ER)-positive or progesterone receptor (PR)-positive breast cancer with ER or PR Allred Score > 4
* Patient must have an ECOG Performance Status of 0-2
* Patients must be able to swallow and retain oral medication

Exclusion Criteria:

* Patient must not have received any prior chemotherapy, radiation therapy, or biologic therapy for invasive breast cancer within the past five years
* Patient must not be pregnant or nursing
* Patient must not have had any prior malignancy except for adequately treated basal cell (or squamous cell) skin cancer, in situ cervical cancer or other cancer for which the patient has been disease-free for five years.
* Women of childbearing age unable or unwilling to use contraception

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laila Agrawal, MD, Principal Investigator — Vanderbilt University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tamoxifen
Started | 35
Completed | 31
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Tamoxifen
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 12
Age, Continuous [Mean (Full Range); unit: years] | 59.1 [35 to 78]
Gender [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Region of Enrollment [Number; unit: participants]
  Guatemala | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Successfully Accrued in the Study, as a Measure of Feasibility
Description: Feasibility is defined as the ability to recruit the stated number of patients and fifty percent of participants completing the trial. Completing the trial is defined as reaching surgery if they are a responder to tamoxifen or obtaining the six week biopsy specimen if they are a non-responder.
Time Frame: 4-6 months
Population: The number of patients analyzed was the accrual goal for number of participants and the outcome measure was the actual number of participants accrued. The outcome measure time frame is the maximum time each participant would be on study.
Measure: Number; unit: participants
Arm/Group | Tamoxifen
Number analyzed (Participants) | 50
participants | 35

2. Secondary Outcome: Number of Participants With Definitive Surgery in Responders to Neoadjuvant Tamoxifen
Description: Rate of definitive surgery after 4 months of neoadjuvant tamoxifen therapy in patients who were deemed to be "responders" to neoadjuvant tamoxifen (Ki67 < or = 10% after 4-6 weeks on neoadjuvant tamoxifen therapy)
Time Frame: 4-6 months
Measure: Number; unit: participants
Arm/Group | Tamoxifen
Number analyzed (Participants) | 35
participants | 13

3. Secondary Outcome: Ki67 Suppression Rate at 4-6 Weeks in Patients Who Underwent an On-treatment Biopsy
Description: Result is the number of participants who had Ki67 suppression (< or = 10%) after 4-6 weeks of neoadjuvant tamoxifen out of patients who underwent an on-treatment biopsy.
Time Frame: 4-6 weeks
Population: 32 of the 35 patients underwent an on-treatment biopsy; 3 patients did not follow-up and were not included in the number of participants analyzed for this measure.
Measure: Number; unit: participants
Arm/Group | Tamoxifen
Number analyzed (Participants) | 32
participants | 15

4. Secondary Outcome: Overall Clinical Response Rate
Description: Clinical response rate was assessed by palpation after 4 months of tamoxifen. Complete response was defined as no palpable primary tumor on clinical examination and lymph nodes < 10 mm. Partial response was defined as at least 30% decrease in the sum of the diameters compared to baseline sum of diameters. The overall clinical response was the sum of the complete clinical response and partial clinical response.
Time Frame: 4-6 months
Population: This Outcome Measure was only assessed among patients undergoing surgery and is a unique outcome measure.
Measure: Number; unit: participants
Arm/Group | Tamoxifen
Number analyzed (Participants) | 13
participants | 13

5. Secondary Outcome: Pathologic Complete Response
Description: Pathologic complete response was defined as no residual tumor at the primary site or the axillary lymph nodes at the time of surgery.
Time Frame: 4-6 months
Population: This Outcome Measure was only assessed among patients who had undergone surgery.
Measure: Number; unit: participants
Arm/Group | Tamoxifen
Number analyzed (Participants) | 13
participants | 1

6. Secondary Outcome: Breast Conserving Therapy
Description: The rate of breast conservation surgery (as opposed to mastectomy) after 4 months of neoadjuvant tamoxifen therapy in patients who were deemed to be "responders" to neoadjuvant tamoxifen (Ki67 < or = 10% after 4-6 weeks on neoadjuvant tamoxifen therapy).
Time Frame: 4-6 months
Population: This outcome measure was analyzed in patients who were treated with 4 months of neoadjuvant tamoxifen
Measure: Number; unit: participants
Arm/Group | Tamoxifen
Number analyzed (Participants) | 15
participants | 0

ADVERSE EVENTS:
Time Frame: 4 weeks - 6 months (time on tamoxifen prior to surgery)
Arm/Group | Tamoxifen
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No